CLINICAL TRIAL: NCT07130916
Title: A Phase 1, Open-Label, Multiple-Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Aumolertinib in European Participants With Locally Advanced or Metastatic, EGFR-mutated Non-Small Cell Lung Cancer
Brief Title: A Study of Aumolertinib in European Participants With Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HS-10296-108
Record Dates: First submitted 2025-07-31; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-10296(Aumolertinib) (Experimental): In Part A, participants will receive aumolertinib 110 mg (2 × 55 mg tablet) once daily, orally administrated under fasted condition (fasting from 2 hours before to 1 hour after dosing) in 21-day treatment cycles. In Part B (i.e., Day 3 of treatment Cycle 2, and beyond), participants may continue study intervention until PD, death, intolerable toxicity, Investigator's decision, lost of follow-up, receiving another anti-cancer therapy, or any other pre-defined discontinuation criteria.
  Interventions: Drug: Aumolertinib

INTERVENTIONS:
Drug: Aumolertinib — In Part A, participants will receive aumolertinib 110 mg (2 × 55 mg tablet) once daily, orally administrated under fasted condition (fasting from 2 hours before to 1 hour after dosing) in 21-day treatment cycles. In Part B, participants may continue study intervention (aumolertinib 110 mg once daily) until PD, death, intolerable toxicity, Investigator's decision, lost of follow-up, receiving another anti-cancer therapy, or any other pre-defined discontinuation criteria.
  Other Names: HS-10296

SUMMARY:
This is a Phase 1, open-label, multicenter, multiple-dose study to evaluate aumolertinib in European participants with a confirmed diagnosis of activating EGFR mutation positive (EGFRm+) locally advanced or metastatic NSCLC.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the PK profile, safety, and tolerability of aumolertinib in European participants with locally advanced or metastatic NSCLC harboring at least one of the EGFR mutations (ex19del, L858R, or T790M). All enrolled participants will receive the study intervention at selected oral dose(s) once daily throughout 21 day cycles. Study details include:

Part A:

During study Part A, participants will be required to present at the study site for PK assessments on Days 1, 2, 8, and 15 of treatment Cycle 1, and on Days 1 and 2 of treatment Cycle 2. Part A will undergo safety assessments and will characterize the PK of aumolertinib and related metabolites following single and multiple doses.

PK samples are to be collected pre-dose (within 1 hour prior to dosing) of treatment with aumolertinib on Days 8 and 15 of treatment Cycle 1, and on Day 1 of treatment Cycles 1 and 2 at the following timepoints: pre-dose (within 1 hour prior to dosing) and 1-, 2-, 3-, 4-, 5-, 6-, 8-, 10 , 12-, and 24-hour (Day 2) post-dose.

Part B:

During Part B of the study (i.e., Day 3 of treatment Cycle 2, and beyond), participants may continue study intervention until PD, death, intolerable toxicity, Investigator's decision, lost of follow-up, receiving another anti-cancer therapy, or any other pre-defined discontinuation criteria. Participants will undergo safety assessments and tumor evaluation according to clinical indication.

The End of Treatment Visit will be conducted within 7 days after determining the participants' discontinuation of the study intervention. The Safety Follow-up (SFU) Visit will be conducted 28 (± 7) days after the last dose of study intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female European participants (inhabitant of a European country and of European descent) must be ≥ 18 years of age, at the time of signing the informed consent.
2. Histological or cytological confirmation diagnosis of newly diagnosed locally advanced (clinical stage IIIB or IIIC) or metastatic (clinical stage IVA or IVB) NSCLC or recurrent NSCLC (per The Eighth Edition of The American Joint Committee on Cancer [AJCC] Cancer Staging Manual in Lung Cancer), not amenable to curative surgery or definitive radiotherapy with or without chemotherapy.

   NOTE: if small cell elements are present, the participant is ineligible.
3. Prior anti-tumor systemic therapy. Participant must fulfill one of below:

   1. Participants who have not received any prior anti-tumor systemic therapy, and the tumor must harbor at least one of the EGFR mutations (ex19del or L858R).
   2. Participants who have received prior neoadjuvant, adjuvant therapies with curative intent for nonmetastatic disease must have completed treatment for at least 12 months prior to the development of recurrent or metastatic disease, and the tumor must harbor at least one of the EGFR mutations (ex19del or L858R).
   3. Participant who only received one line of first- or second-generation EGFR-TKI in the locally advanced or metastatic setting and have documented radiological progression prior to enrolling in the study, and the tumor must harbor EGFR T790M mutation.
4. Confirmation that the tumor harbors at least one of the EGFR mutations (ex19del, L858R, or T790M) using a clinically validated assay in a licensed laboratory with applicable local accreditation based on tumor tissue and/or circulating tumor deoxyribonucleic acid (ctDNA) in blood.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-1 and no deterioration in the previous two weeks with a minimum life expectancy of 12 weeks.
6. Participants must have evaluable disease. At least one measurable (not previously irradiated) and/or non-measurable lesions per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (Appendix 6) that can be accurately assessed at baseline and suitable for repeated assessments by computed tomography (CT) or magnetic resonance imaging (MRI) scans. If only one measurable lesion exists, it is acceptable to be used (as a target lesion [TL]) as long as it has not been previously irradiated and as long as it has not been biopsied within 14 days of the baseline tumor assessment scans.
7. Adequate bone marrow reserve or organ function without blood transfusion or growth factor support ≤ 14 days before sample collection at screening as demonstrated by any of the following laboratory values:

   1. Absolute neutrophil count ≥ 1.5 × 109/L;
   2. Platelet count ≥ 80 × 109/L;
   3. Hemoglobin ≥ 90 g/L;
   4. ALT ≤ 2.5 × upper limit of normal (ULN) if no demonstrable liver metastases or ≤ 5 × ULN in the presence of liver metastases;
   5. AST ≤ 2.5 × ULN if no demonstrable liver metastases or ≤ 5 × ULN in the presence of liver metastases;
   6. Total bilirubin (TBL) ≤ 1.5 × ULN if no liver metastases or ≤ 3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia) or liver metastases;
   7. Creatinine ≤ 1.5 × ULN concurrent with creatinine clearance ≥ 50 mL/min (measured or calculated by Cockcroft and Gault equation);
   8. The confirmation of creatinine clearance is only required when creatinine is ≤ 1.5 × ULN;
   9. International normalized ratio (INR) ≤ 1.5;
   10. Activated partial thromboplastin time ≤ 1.5 ULN;
8. Contraceptive use by men and women must be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   NOTE: The reliability of sexual abstinence for male and/or female enrollment eligibility needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post ovulation methods) and withdrawal are not acceptable methods of contraception.

   Male Participants:

   • A male participant must agree to use a highly effective contraception as detailed in Appendix 4 of this protocol from screening to three months after the last dose of study intervention.

   Female Participants:

   • A female participant is eligible to participate if she has a negative pregnancy test no later than 72 hours prior to start of dosing if of childbearing potential, not breastfeeding from screening to three months after the last dose of the study intervention, and at least one of the following conditions applies:
   * Not a woman of childbearing potential (WOCBP) as defined in Appendix 4. OR
   * A WOCBP who agrees to follow the contraceptive guidance in Appendix 4 from screening to three months after the last dose of study intervention and should not be breastfeeding from screening to three months after the last dose of the study intervention.
9. Participant is capable of giving signed informed consent as described in Appendix 1, Section 10.1.3 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study intervention with the exception of alopecia and Grade 2 neurotoxicity related to prior platinum-therapy.
2. History of another primary malignancy except for the malignancy treated with curative intent with no known active disease ≤ 5 years before the first dose of study intervention and of low potential risk for recurrence. Exceptions include, but are not limited to, adequately resected non melanoma skin cancer, and curatively treated in situ disease.
3. Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids for at least four weeks prior to start of study intervention.
4. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding within two weeks prior to the first dose of study intervention, active infection (e.g., active HBV infection, HCV infection), or HIV infection, which in the Investigator's opinion makes it undesirable for the participant to participate in the study or which would jeopardise compliance with the protocol.
5. Any of the following cardiac criteria: mean resting corrected QT (QT; the time from the start of the Q wave to the end of the T wave in an ECG) interval corrected for heart rate using Fridericia's correction factor (QTcF) > 470 ms obtained from three ECGs; any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g., complete left bundle branch block, third degree heart block, second degree heart block, PR interval > 250 ms; any factors that increase the risk of corrected QT (QTc) prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under age of 40 or any concomitant medication known to prolong the QT interval; Left ventricular ejection fraction (LVEF) ≤ 40%.
6. Past medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
7. Refractory nausea, vomiting, or chronic GI disorders; Participants unable to swallow oral medication or participants with GI disorders or significant GI resection likely to interfere with the absorption of study intervention.
8. Participant has any disease or condition that, in the judgment of the physician, may increase the risk to the safety or interfering with study assessments.
9. Participant with a known hypersensitivity to study intervention, structural analog, or any of the excipients of the products.
10. Received any of the following treatments:

    1. Treatment with a first- or second-generation EGFR-TKI (e.g., erlotinib or gefitinib) within 8 days of the first dose of study intervention or 5 half-lives, whichever is the longer.
    2. Treatment with prior third-generation EGFR-TKI (e.g., osimertinib).
    3. Any cytotoxic chemotherapy, investigational agents or other anticancer drugs from a previous treatment regimen or clinical study taken within 14 days of the first dose of study intervention or 5 half lives, whichever is longer.
    4. Treatment with medications known to be potent strong inhibitors or inducers of CYP3A4 or narrow therapeutic index drugs for CYP3A4 sensitive substrates (see Appendix 7) within 7 days of the first dose of study intervention or 5 half-lives, whichever is the longer.
    5. Major surgery (excluding placement of vascular access) within four weeks of the first dose of study intervention.
    6. Radiotherapy with a limited field of radiation for palliation within one week prior to the first dose of study intervention or receiving radiation with more than 30% of the bone marrow or with a wide field of radiation within four weeks prior to the first dose of study intervention.
11. Participants participated in any interventional clinical study or had been treated with any investigational drugs within 28 days or 5 half-lives, whichever is longer, before Screening Visit.

    Other Exclusion Criteria
12. Participant who, in the judgment of the Investigator, may have poor compliance with the procedures, limitations, and requirements of the study and are not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-08-09 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Tmax of of single and multiple doses of aumolertinib, its metabolite HAS-719, and other related metabolites in European participants with locally advanced or metastatic, epidermal growth factor receptor (EGFR)-mutated non-small cell lung cancer (NSCLC). | Cycle2 Day1（each cycle is 21 days）
  Time to reach Cmax
Cmax of of single and multiple doses of aumolertinib, its metabolite HAS-719, and other related metabolites in European participants with locally advanced or metastatic, epidermal growth factor receptor (EGFR)-mutated non-small cell lung cancer (NSCLC). | Cycle2 Day1（each cycle is 21 days）
  Maximum plasma concentration
AUC0-24h of of single and multiple doses of aumolertinib, its metabolite HAS-719, and other related metabolites in European participants with locally advanced or metastatic, epidermal growth factor receptor (EGFR)-mutated non-small cell lung cancer | Cycle2 Day1（each cycle is 21 days）
  Area under the plasma concentration-time curve form 0-24h
Cmin of of single and multiple doses of aumolertinib, its metabolite HAS-719, and other related metabolites in European participants with locally advanced or metastatic, epidermal growth factor receptor (EGFR)-mutated non-small cell lung cancer (NSCLC). | Cycle2 Day1（each cycle is 21 days）
  Minmum plasma concentration

SECONDARY OUTCOMES:
Adverse events (AEs) of aumolertinib administered in European participants with locally advanced or metastatic, EGFR-mutated NSCLC. | Through study completion, an average of 18 months
  Incidence and severity of advese event

CONTACTS AND LOCATIONS:
Locations (6):
- Bosnia and Herzegovina (4):
  - Republika Srpska University Clinical Centre of the Republic of Srpska, Dvanaest beba bb, Banja Luka
  - University Clinical Hospital Mosta, Bijeli Brijeg bb, Mostar
  - Clinical Center University of Sarajevo, Bolnicka 25, Sarajevo
  - Cantonal Hospital Zenica, Crkvice 67, Zenica
- MHAT "Sveta Sofia" Departmet of Medical Oncology Bulgaria Blvd, Sofia, Grad, Bulgaria
- Arensia Exploratory Medicine Moldova - IMSP Institutul Oncologic. Strada Nicolae Testemitanu Nr 30, Chisinau, Moldova